CLINICAL TRIAL: NCT01090362
Title: Prospective, Multi Centre, International Registry of Male and Female Patients Newly Diagnosed With Atrial Fibrillation.
Brief Title: Global Anticoagulant Registry in the Field
Acronym: GARFIELD-AF
Status: Completed | Type: Observational
Sponsor: Thrombosis Research Institute (Other)
Collaborators: Bayer (Industry); University of Birmingham (Other); Brigham and Women's Hospital (Other); Quintiles, Inc. (Industry); Advanced Drug and Device Services SAS (Unknown); Apothecaries Clinical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: TRI08888
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Anticoagulation; Stroke; Stroke prevention; Health Economics
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Cohort 1: Cohort complete with 5,088 retrospective patients and 5,499 prospective patients recruited from 19 countries.
- Cohort 2: Cohort completed with 11,351 patients enrolled from 30 countries
- Cohort 3: Cohort 3 completed with 11,139 patients enrolled globally from 32 countries
- Cohort 4: Cohort 4 completed with 11,2780 patients enrolled from 35 countries.
- Cohort 5: Final cohort completed with 12,186 patients enrolled.

SUMMARY:
The Global Anticoagulant Registry in the FIELD-Atrial Fibrillation (GARFIELD-AF Registry) is a non-interventional, observational study that characterized a global population of non-valvular atrial fibrillation patients. The registry was used to document global baseline characteristics, current treatment strategies and outcome measures. Characterisation of a number of AF sub-populations was also completed. GARFIELD-AF is an independent academic research initiative sponsored by the Thrombosis Research Institute (London, UK) and supported by an unrestricted research grant from Bayer AG (Berlin, Germany).

DETAILED DESCRIPTION:
Using data from more than 1000 randomly selected centres across 35 countries, representing all possible care settings, the registry will help to characterize real-life anticoagulant treatment patterns and outcomes, including rates of stroke and bleeding complications, as well as provide data on other important issues, such as physicians' compliance with guidelines and patients' adherence to therapy. This is particularly timely as standard practice moves away from vitamin K antagonist (VKA)-dominated therapy and towards a new era of novel oral anticoagulants (OACs), i.e. direct Factor Xa inhibitors and direct thrombin inhibitors.

To ensure a dataset that truly reflects current practice, the investigators are requested to prospectively enrol all newly diagnosed patients with non-valvular AF who have at least one additional investigator-determined risk factor for stroke. Patients are consecutively recruited into one of five cohorts and followed up for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

Prospective Cohort

* Written informed consent
* Age 18 years and older
* New diagnosis of non-valvular atrial fibrillation (diagnosed within the last 6 weeks) with at least one additional risk factor for stroke and regardless of therapy.

Retrospective validation cohort

* Written informed consent
* Age 18 years and older
* Diagnosis of non-valvular AF (diagnosed 6-24 months prior to enrolment) with at least one additional risk factor for stroke and regardless of therapy.

Exclusion criteria:

* No further follow-up envisaged or possible within enrolling hospital or with associated family practitioner.
* Patients with transient AF secondary to a reversible cause.
* Patients recruited in controlled clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients newly diagnosed with atrial fibrillation (AF) who are with at least one additional risk of stroke from 18 countries globally.
Sampling Method: Non-Probability Sample
Enrollment: 57250 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Death | 4 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 8 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 12 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 16 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 20 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 24 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 3 years
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 4 years
  All cause mortality including cardiovascular and non-cardiovascular death
Stroke/Systemic embolism (SE) | 4 months
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 8 months
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 12 months
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 16 months
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 20 months
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 24 months
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 3 years
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Stroke/Systemic embolism (SE) | 4 years
  Stroke/SE was defined as the combined end points of ischemic stroke, and SE
Major bleeding | 4 months
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 8 months
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 12 months
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 16 months
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 20 months
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 24 months
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 3 years
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.
Major bleeding | 4 years
  Defined as clinically overt bleeding associated with a critical site or hemorrhagic stroke, a fall in haemoglobin of ≥2 g/dl, transfusion of ≥2 units of packed red blood cells, or fatal outcome.

SECONDARY OUTCOMES:
Cerebrovascular events defined as Stroke | 4 months
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 8 months
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 12 months
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 16 months
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 20 months
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 24 months
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 3 years
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Cerebrovascular events defined as Stroke | 4 years
  Primary ischaemic stroke, Primary intracerebral haemorrhage, Secondary haemorrhagic ischaemic stroke.
Transient Ischemic Attacks (TIA) | 4 months
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 8 months
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 12 months
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 16 months
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 20 months
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 24 months
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 3 years
  Number of Transient Ischemic Attacks (TIA)
Transient Ischemic Attacks (TIA) | 4 years
  Number of Transient Ischemic Attacks (TIA)
Acute coronary syndromes | 4 months
  Number including unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 8 months
  Number including unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 12 months
  Number Including unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 16 months
  Number including unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 20 months
  Number including unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 24 months
  Number including Unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 3 years
  Number including unstable angina, STEMI, Non-STEMI
Acute coronary syndromes | 4 years
  Number including unstable angina, STEMI, Non-STEMI
Therapy persistence | 4 months
  Participant duration of time on therapy
Therapy persistence | 8 months
  Participant duration of time on therapy
Therapy persistence | 12 months
  Participant duration of time on therapy
Therapy persistence | 16 months
  Participant duration of time on therapy
Therapy persistence | 20 months
  Participant duration of time on therapy
Therapy persistence | 24 months
  Participant duration of time on therapy
Therapy persistence | 3 years
  Participant rate of discontinuation
Therapy persistence | 4 years
  Participant duration of time on therapy
Incidences of other clinical events | 4 months
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 8 months
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 12 months
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 16 months
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 20 months
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 24 months
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 3 years
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Incidences of other clinical events | 4 years
  Myocardial infarction (MI)/ acute coronary syndromes (ACS), and congestive heart failure (CHF)
Bleeding Events | 4 months
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 8 months
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 12 months
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 16 months
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 20 months
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 24 months
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 3 years
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Bleeding Events | 4 years
  Frequency, severity, location, outcome, Healthcare utilisation used for bleeding event
Pulmonary Embolism | 4 months
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 8 months
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 12 months
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 16 months
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 20 months
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 24 months
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 3 years
  Number of participants with a Pulmonary Embolism
Pulmonary Embolism | 4 years
  Number of participants with a Pulmonary Embolism

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Kakkar, Study Director — Thrombosis Research Institute, London, UK
Locations (35):
- Prof. Samuel Goldhaber, Boston, Massachusetts, United States
- Dr Hector Luciardi, National Co-ordinating Investigator, National University of Tucuman, San Miguel de Tucumán, Argentina
- Harry Gibbs, National Co-ordinating Investigator, The Alfred Hospital, Melbourne, Australia
- Marianne Brodmann: National Co-ordinating Investigator, Medizinische Universität Graz, Graz, Austria
- Dr Frank Cools, National Co-ordinating Investigator, AZ Klina, Brasschaat, Belgium
- Dr Antonio Barretto, National Coordinating Investigator, Hospital Santa Marcelina,, São Paulo, Brazil
- Prof Stuart Connolly and Dr John Eikelboom, National Coodinating Investigators, Mc Master University, Hamilton, Canada
- Dr Ramon Corbalan, National Coordinating Investigator, Pontifica Universidad Catolica de Chile, Santiago, Chile
- Prof Zin-Cheng, National Coordinating Investigator, Peking Union Medical College & Chinese Academy Medical Sciences People Hospital, Beijing, China
- Dr Petr Jansky, National Coordinating Investigator, Cardiovaskular Center, Motol Univesity Hospital, Prague, Czechia
- Prof Joern Dalsgaard Nielsen, National Coordinating Investigator, Bispebjerg & Frederiksberg Hospitals, Frederiksberg, Denmark
- Dr. Hany Ragy, National Coordinating Investigator, Hayat Hospital, Cairo, Egypt
- Prof Pekka Raatikainen, National Coordinating Investigator, Univesrsity of Tampere, Tampere, Finland
- Prof. Jean-Yues LeHeuzey, National Coordinating Investigator, Hopital Europeen Georges Pompidou, Paris, France
- Prof Harald Darius, National oordinating Investigator, Vivantes Klinikum Neukölln, Berlin, Germany
- Dr Matyas Keltai, National Coordinating Investigator, Hungarian Institute of Cardiology, Budapest, Hungary
- Dr Sawney, National Coordinating Investigator, Sir Ganga Ram Hospital, New Delhi, Bangalore, India
- Profs Giancarlo Agnelli and Giuseppe Ambrosio, National Coordinating Investigators, University of Perugia, Perugia, Italy
- Professor Yukihiro Koretsune, National Coordinating Investigator, Osaka National Hospital, Osaka, Japan
- Dr Carlos Jerjes Sanchez Diaz, National Coordinating Investigator,Tecnologico de Monterrey, Monterrey, Mexico
- Professor Hugo ten Cate, National Coordinating Investigator, Cardiovascular Research Institute Maastricht, Maastricht, Netherlands
- Professor Dan Atar, National Coordinating Investigator, Oslo University Hospital, Oslo, Norway
- Prof Janina Stępińska, National Coordinating Investigator, Institute of Cardiology, Warsaw, Warsaw, Poland
- Professor Elizaveta Panchenko, National Coordinating Investigator, Cardiology Research and Production Center, Moscow, Russia
- Dr Toon Wei Lim, National Coordinating Investigator, National University Hospital, Singapore, Singapore
- Prof. Barry Jacobson, National Coordinating Investigator, University of the Witwatersrand, Johannesburg, South Africa
- Prof. Seil Oh, National Coordinating Investigator, National University Hospital, Seoul, South Korea
- Dr Xavier Vinolas, National Coordinating Investigator, Hospital Santa Creu y San Pau, Barcelona, Spain
- Dr Marten Rosenqvist, National Coordinating Investigator, Karolinska Institute, Stockholm, Sweden
- Dr Jan Steffel, National Coordinating Investigator, University Hospital, Zurich, Switzerland
- Prof. Pantep Angchaisuksiri, National Coordinating Investigator, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand
- Professor Ali Oto, National Coordinating Investigator, Memorial Ankara Hospital, Ankara, Turkey (Türkiye)
- Prof. Alexandr Parkhomenko, National Coordinating Investigator, Strazhesko Institute of Cardiology, Kiev, Ukraine
- Prof. Wael Al Mahmeed, National Coordinating Investigator, SKMC Cardiac Siences, Abu Dhabi, United Arab Emirates
- Prof. David Fitzmaurice, National Coordinating Investigator, University of Warwick, Coventry, United Kingdom

REFERENCES:
- [Background] Kakkar AK, Mueller I, Bassand JP, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Hacke W, Lip GY, Mantovani LG, Verheugt FW, Jamal W, Misselwitz F, Rushton-Smith S, Turpie AG. International longitudinal registry of patients with atrial fibrillation at risk of stroke: Global Anticoagulant Registry in the FIELD (GARFIELD). Am Heart J. 2012 Jan;163(1):13-19.e1. doi: 10.1016/j.ahj.2011.09.011. Epub 2011 Nov 20. PMID 22172431
- [Background] Apenteng PN, Murray ET, Holder R, Hobbs FD, Fitzmaurice DA; UK GARFIELD Investigators and GARFIELD Steering Committee. An international longitudinal registry of patients with atrial fibrillation at risk of stroke (GARFIELD): the UK protocol. BMC Cardiovasc Disord. 2013 Apr 23;13:31. doi: 10.1186/1471-2261-13-31. PMID 23617744
- [Background] Aalbers J. GARFIELD: a window on the real-life treatment of atrial fibrillation - South Africa joins the GARFIELD registry. Cardiovasc J Afr. 2012 Oct;23(9):528. No abstract available. PMID 23108524
- [Result] Kakkar AK, Mueller I, Bassand JP, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Hacke W, Lip GY, Mantovani LG, Turpie AG, van Eickels M, Misselwitz F, Rushton-Smith S, Kayani G, Wilkinson P, Verheugt FW; GARFIELD Registry Investigators. Risk profiles and antithrombotic treatment of patients newly diagnosed with atrial fibrillation at risk of stroke: perspectives from the international, observational, prospective GARFIELD registry. PLoS One. 2013 May 21;8(5):e63479. doi: 10.1371/journal.pone.0063479. Print 2013. PMID 23704912
- [Derived] Cheng CY, Lian TY, Zhu XJ, Virdone S, Sun K, Camm J, Li XM, Goto S, Pieper K, Kayani G, Fang XH, Jing ZC, Kakkar AK; GARFIELD-AF Investigators. Atrial fibrillation outcomes in patients from Asia and non-Asia countries: insights from GARFIELD-AF. Open Heart. 2025 Feb 6;12(1):e003109. doi: 10.1136/openhrt-2024-003109. PMID 39914996
- [Derived] Himmelreich JCL, Virdone S, Camm AJ, Pieper K, Harskamp RE, Verheugt FWA, Bassand JP, Misselwitz F, Pereira-Barretto AC, Cools F, Gibbs H, Kakkar AK; GARFIELD-AF investigators. Emulation of ARISTOTLE and ROCKET AF trials in real-world atrial fibrillation patients results in similar efficacy and safety as original landmark trials: insights from the GARFIELD-AF registry. Open Heart. 2025 Jan 19;12(1):e002966. doi: 10.1136/openhrt-2024-002966. PMID 39832940
- [Derived] Camm CF, Virdone S, Jerjes-Sanchez C, Oh S, Eikelboom JW, Oto A, Fox KAA, Camm AJ, Pieper KS, Goto S, Ragy H, Kakkar AK; GARFIELD-AF registry. Association of care specialty with anticoagulant prescription and clinical outcomes in newly diagnosed atrial fibrillation: Results from the GARFIELD-AF registry. Int J Cardiol. 2025 Feb 15;421:132866. doi: 10.1016/j.ijcard.2024.132866. Epub 2024 Dec 2. PMID 39631531
- [Derived] Bassand JP, Virdone S, Camm AJ, Fox KAA, Goldhaber SZ, Goto S, Haas S, Hacke W, Kayani G, Keltai M, Misselwitz F, Pieper KS, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Oral anticoagulation across diabetic subtypes in patients with newly diagnosed atrial fibrillation: A report from the GARFIELD-AF registry. Diabetes Obes Metab. 2023 Oct;25(10):3040-3053. doi: 10.1111/dom.15202. Epub 2023 Jul 12. PMID 37435777
- [Derived] Camm AJ, Steffel J, Virdone S, Bassand JP, Fox KAA, Goldhaber SZ, Goto S, Haas S, Turpie AGG, Verheugt FWA, Misselwitz F, Herreros RC, Kayani G, Pieper KS, Kakkar AK; GARFIELD-AF Investigators. Guideline-directed medical therapies for comorbidities among patients with atrial fibrillation: results from GARFIELD-AF. Eur Heart J Open. 2023 May 19;3(3):oead051. doi: 10.1093/ehjopen/oead051. eCollection 2023 May. PMID 37293139
- [Derived] Yuan L, Yang L, Zhang S, Xu Z, Qin J, Shi Y, Yu P, Wang Y, Bao Z, Xia Y, Sun J, He W, Chen T, Chen X, Hu C, Zhang Y, Dong C, Zhao P, Wang Y, Jiang N, Lv B, Xue Y, Jiao B, Gao H, Chai K, Li J, Wang H, Wang X, Guan X, Liu X, Zhao G, Zheng Z, Yan J, Yu H, Chen L, Ye Z, You H, Bao Y, Cheng X, Zhao P, Wang L, Zeng W, Tian Y, Chen M, You Y, Yuan G, Ruan H, Gao X, Xu J, Xu H, Du L, Zhang S, Fu H, Cheng X. Development of a tongue image-based machine learning tool for the diagnosis of gastric cancer: a prospective multicentre clinical cohort study. EClinicalMedicine. 2023 Feb 6;57:101834. doi: 10.1016/j.eclinm.2023.101834. eCollection 2023 Mar. PMID 36825238
- [Derived] van Husen G, Virdone S, Pieper K, Kayani G, Fox KAA. Universal Clinician Device for improving risk prediction and management of patients with atrial fibrillation: an assumed benefit analysis. Eur Heart J Digit Health. 2022 Mar 25;3(2):181-194. doi: 10.1093/ehjdh/ztac011. eCollection 2022 Jun. PMID 36713019
- [Derived] Fox KAA, Virdone S, Bassand JP, Camm AJ, Goto S, Goldhaber SZ, Haas S, Kayani G, Koretsune Y, Misselwitz F, Oh S, Piccini JP, Parkhomenko A, Sawhney JPS, Stepinska J, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF investigators*. Do baseline characteristics and treatments account for geographical disparities in the outcomes of patients with newly diagnosed atrial fibrillation? The prospective GARFIELD-AF registry. BMJ Open. 2022 Jan 7;12(1):e049933. doi: 10.1136/bmjopen-2021-049933. PMID 34996784
- [Derived] Pope MK, Hall TS, Schirripa V, Radic P, Virdone S, Pieper KS, Le Heuzey JY, Jansky P, Fitzmaurice DA, Cappato R, Atar D, Camm AJ, Kakkar AK; GARFIELD-AF investigators. Cardioversion in patients with newly diagnosed non-valvular atrial fibrillation: observational study using prospectively collected registry data. BMJ. 2021 Oct 27;375:e066450. doi: 10.1136/bmj-2021-066450. PMID 34706884
- [Derived] Cools F, Johnson D, Camm AJ, Bassand JP, Verheugt FWA, Yang S, Tsiatis A, Fitzmaurice DA, Goldhaber SZ, Kayani G, Goto S, Haas S, Misselwitz F, Turpie AGG, Fox KAA, Pieper KS, Kakkar AK; GARFIELD-AF Investigators. Risks associated with discontinuation of oral anticoagulation in newly diagnosed patients with atrial fibrillation: Results from the GARFIELD-AF Registry. J Thromb Haemost. 2021 Sep;19(9):2322-2334. doi: 10.1111/jth.15415. Epub 2021 Jul 23. PMID 34060704
- [Derived] Fox KAA, Virdone S, Pieper KS, Bassand JP, Camm AJ, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Kayani G, Oto A, Misselwitz F, Piccini JP, Dalgaard F, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. GARFIELD-AF risk score for mortality, stroke, and bleeding within 2 years in patients with atrial fibrillation. Eur Heart J Qual Care Clin Outcomes. 2022 Mar 2;8(2):214-227. doi: 10.1093/ehjqcco/qcab028. PMID 33892489
- [Derived] Pope MK, Atar D, Svilaas A, Hole T, Nielsen JD, Hintze U, Crisby M, Raatikainen P, Airaksinen KEJ, Virdone S, Pieper K, Kayani G, Le Heuzey JY, Steffel J, Stepinska J, Bassand JP, Camm AJ; GARFIELD-AF Investigators. Risk profile, antithrombotic treatment and clinical outcomes of patients in Nordic countries with atrial fibrillation - results from the GARFIELD-AF registry. Ann Med. 2021 Dec;53(1):485-494. doi: 10.1080/07853890.2021.1893897. PMID 33818226
- [Derived] Sayin BY, Al Mahmeed W, Ragy HI, Elbahry A, Virdone S, Kakkar AK, Ersanli M, Oto A. Middle East Treatment Strategies and Clinical Outcomes in Patients with Atrial Fibrillation: One-Year Follow-up Data from Garfield-AF Study. Adv Ther. 2021 May;38(5):2391-2405. doi: 10.1007/s12325-021-01670-5. Epub 2021 Mar 27. PMID 33772428
- [Derived] Gibbs H, Freedman B, Rosenqvist M, Virdone S, Mahmeed WA, Ambrosio G, Camm AJ, Jacobson B, Jerjes-Sanchez C, Kayani G, Oto A, Panchenko E, Ragy H, Kakkar AK; GARFIELD-AF Investigators. Clinical Outcomes in Asymptomatic and Symptomatic Atrial Fibrillation Presentations in GARFIELD-AF: Implications for AF Screening. Am J Med. 2021 Jul;134(7):893-901.e11. doi: 10.1016/j.amjmed.2021.01.017. Epub 2021 Feb 16. PMID 33607088
- [Derived] Bassand JP, Virdone S, Badoz M, Verheugt FWA, Camm AJ, Cools F, Fox KAA, Goldhaber SZ, Goto S, Haas S, Hacke W, Kayani G, Misselwitz F, Pieper KS, Turpie AGG, van Eickels M, Kakkar AK. Bleeding and related mortality with NOACs and VKAs in newly diagnosed atrial fibrillation: results from the GARFIELD-AF registry. Blood Adv. 2021 Feb 23;5(4):1081-1091. doi: 10.1182/bloodadvances.2020003560. PMID 33606006
- [Derived] Camm AJ, Fox KAA, Virdone S, Bassand JP, Fitzmaurice DA, Berchuck SI, Gersh BJ, Goldhaber SZ, Goto S, Haas S, Misselwitz F, Pieper KS, Turpie AGG, Verheugt FWA, Cappato R, Kakkar AK; GARFIELD-AF investigators. Comparative effectiveness of oral anticoagulants in everyday practice. Heart. 2021 May 26;107(12):962-970. doi: 10.1136/heartjnl-2020-318420. PMID 33593994
- [Derived] Camm AJ, Cools F, Virdone S, Bassand JP, Fitzmaurice DA, Arthur Fox KA, Goldhaber SZ, Goto S, Haas S, Mantovani LG, Kayani G, Grierson Turpie AG, Antoon Verheugt FW, Kakkar AK; GARFIELD-AF Investigators. Mortality in Patients With Atrial Fibrillation Receiving Nonrecommended Doses of Direct Oral Anticoagulants. J Am Coll Cardiol. 2020 Sep 22;76(12):1425-1436. doi: 10.1016/j.jacc.2020.07.045. PMID 32943160
- [Derived] Bassand JP, Apenteng PN, Atar D, Camm AJ, Cools F, Corbalan R, Fitzmaurice DA, Fox KA, Goto S, Haas S, Hacke W, Jerjes-Sanchez C, Koretsune Y, Heuzey JL, Sawhney JP, Oh S, Stepinska J, Cate VT, Verheugt FW, Kayani G, Pieper KS, Kakkar AK, Garfield-Af Investigators FT. GARFIELD-AF: a worldwide prospective registry of patients with atrial fibrillation at risk of stroke. Future Cardiol. 2021 Jan;17(1):19-38. doi: 10.2217/fca-2020-0014. Epub 2020 Jul 22. PMID 32696663
- [Derived] Hacke W, Bassand JP, Virdone S, Camm AJ, Fitzmaurice DA, Fox KA, Goldhaber SZ, Goto S, Haas S, Kayani G, Mantovani LG, Misselwitz F, Pieper KS, Turpie AG, van Eickels M, Verheugt FW, Kakkar AK; GARFIELD-AF Investigators. Prior stroke and transient ischemic attack as risk factors for subsequent stroke in atrial fibrillation patients: A report from the GARFIELD-AF registry. Int J Stroke. 2020 Apr;15(3):308-317. doi: 10.1177/1747493019891516. Epub 2019 Dec 17. PMID 31847794
- [Derived] Atar D, Berge E, Le Heuzey JY, Virdone S, Camm AJ, Steffel J, Gibbs H, Goldhaber SZ, Goto S, Kayani G, Misselwitz F, Stepinska J, Turpie AGG, Bassand JP, Kakkar AK; GARFIELD-AF Investigators. The association between patterns of atrial fibrillation, anticoagulation, and cardiovascular events. Europace. 2020 Feb 1;22(2):195-204. doi: 10.1093/europace/euz292. PMID 31747004
- [Derived] Verheugt FWA, Ambrosio G, Atar D, Bassand JP, Camm AJ, Costabel JP, Fitzmaurice DA, Illingworth L, Goldhaber SZ, Goto S, Haas S, Jansky P, Kayani G, Stepinska J, Turpie AGG, van Eickels M, Kakkar AK; GARFIELD-AF Investigators. Outcomes in Newly Diagnosed Atrial Fibrillation and History of Acute Coronary Syndromes: Insights from GARFIELD-AF. Am J Med. 2019 Dec;132(12):1431-1440.e7. doi: 10.1016/j.amjmed.2019.06.008. Epub 2019 Jul 12. PMID 31306621
- [Derived] Haas S, Camm AJ, Bassand JP, Angchaisuksiri P, Cools F, Corbalan R, Gibbs H, Jacobson B, Koretsune Y, Mantovani LG, Misselwitz F, Panchenko E, Ragy HI, Stepinska J, Turpie AG, Sawhney JP, Steffel J, Lim TW, Pieper KS, Virdone S, Verheugt FW, Kakkar AK; GARFIELD-AF Investigators. Predictors of NOAC versus VKA use for stroke prevention in patients with newly diagnosed atrial fibrillation: Results from GARFIELD-AF. Am Heart J. 2019 Jul;213:35-46. doi: 10.1016/j.ahj.2019.03.013. Epub 2019 Apr 11. PMID 31128503
- [Derived] Corbalan R, Bassand JP, Illingworth L, Ambrosio G, Camm AJ, Fitzmaurice DA, Fox KAA, Goldhaber SZ, Goto S, Haas S, Kayani G, Mantovani LG, Misselwitz F, Pieper KS, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Analysis of Outcomes in Ischemic vs Nonischemic Cardiomyopathy in Patients With Atrial Fibrillation: A Report From the GARFIELD-AF Registry. JAMA Cardiol. 2019 Jun 1;4(6):526-548. doi: 10.1001/jamacardio.2018.4729. PMID 31066873
- [Derived] Jerjes-Sanchez C, Corbalan R, Barretto ACP, Luciardi HL, Allu J, Illingworth L, Pieper KS, Kayani G; GARFIELD-AF Investigators. Stroke prevention in patients from Latin American countries with non-valvular atrial fibrillation: Insights from the GARFIELD-AF registry. Clin Cardiol. 2019 May;42(5):553-560. doi: 10.1002/clc.23176. Epub 2019 Apr 9. PMID 30873623
- [Derived] Goto S, Angchaisuksiri P, Bassand JP, Camm AJ, Dominguez H, Illingworth L, Gibbs H, Goldhaber SZ, Goto S, Jing ZC, Haas S, Kayani G, Koretsune Y, Lim TW, Oh S, Sawhney JPS, Turpie AGG, van Eickels M, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Management and 1-Year Outcomes of Patients With Newly Diagnosed Atrial Fibrillation and Chronic Kidney Disease: Results From the Prospective GARFIELD - AF Registry. J Am Heart Assoc. 2019 Feb 5;8(3):e010510. doi: 10.1161/JAHA.118.010510. PMID 30717616
- [Derived] Bassand JP, Virdone S, Goldhaber SZ, Camm AJ, Fitzmaurice DA, Fox KAA, Goto S, Haas S, Hacke W, Kayani G, Mantovani LG, Misselwitz F, Pieper KS, Turpie AGG, van Eickels M, Verheugt FWA, Kakkar AK. Early Risks of Death, Stroke/Systemic Embolism, and Major Bleeding in Patients With Newly Diagnosed Atrial Fibrillation. Circulation. 2019 Feb 5;139(6):787-798. doi: 10.1161/CIRCULATIONAHA.118.035012. PMID 30586740
- [Derived] Sawhney JP, Kothiwale VA, Bisne V, Durgaprasad R, Jadhav P, Chopda M, Vanajakshamma V, Meena R, Vijayaraghavan G, Chawla K, Allu J, Pieper KS, John Camm A, Kakkar AK; GARFIELD-AF Investigators. Risk profiles and one-year outcomes of patients with newly diagnosed atrial fibrillation in India: Insights from the GARFIELD-AF Registry. Indian Heart J. 2018 Nov-Dec;70(6):828-835. doi: 10.1016/j.ihj.2018.09.001. Epub 2018 Sep 12. PMID 30580852
- [Derived] Cools F, Wollaert B, Vervoort G, Verstraete S, Voet J, Hermans K, Heyse A, De Wolf A, Hollanders G, Boussy T, Anne W, Vercammen J, Faes D, Beutels M, Mairesse G, Purnode P, Blankoff I, Vandergoten P, Capiau L, Allu J, Bassand JP, Kayani G; GARFIELD-AF Investigators. Treatment patterns in anticoagulant therapy in patients with newly diagnosed atrial fibrillation in Belgium: results from the GARFIELD-AF registry. Acta Cardiol. 2019 Aug;74(4):309-318. doi: 10.1080/00015385.2018.1494089. Epub 2018 Oct 27. PMID 30369290
- [Derived] Bassand JP, Accetta G, Al Mahmeed W, Corbalan R, Eikelboom J, Fitzmaurice DA, Fox KAA, Gao H, Goldhaber SZ, Goto S, Haas S, Kayani G, Pieper K, Turpie AGG, van Eickels M, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Risk factors for death, stroke, and bleeding in 28,628 patients from the GARFIELD-AF registry: Rationale for comprehensive management of atrial fibrillation. PLoS One. 2018 Jan 25;13(1):e0191592. doi: 10.1371/journal.pone.0191592. eCollection 2018. PMID 29370229
- [Derived] Apenteng PN, Gao H, Hobbs FR, Fitzmaurice DA; UK GARFIELD-AF Investigators and GARFIELD-AF Steering Committee. Temporal trends in antithrombotic treatment of real-world UK patients with newly diagnosed atrial fibrillation: findings from the GARFIELD-AF registry. BMJ Open. 2018 Jan 13;8(1):e018905. doi: 10.1136/bmjopen-2017-018905. PMID 29331969
- [Derived] Verheugt FWA, Gao H, Al Mahmeed W, Ambrosio G, Angchaisuksiri P, Atar D, Bassand JP, Camm AJ, Cools F, Eikelboom J, Kayani G, Lim TW, Misselwitz F, Pieper KS, van Eickels M, Kakkar AK; GARFIELD-AF Investigators. Characteristics of patients with atrial fibrillation prescribed antiplatelet monotherapy compared with those on anticoagulants: insights from the GARFIELD-AF registry. Eur Heart J. 2018 Feb 7;39(6):464-473. doi: 10.1093/eurheartj/ehx730. PMID 29281086
- [Derived] Fox KAA, Lucas JE, Pieper KS, Bassand JP, Camm AJ, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Hacke W, Kayani G, Oto A, Mantovani LG, Misselwitz F, Piccini JP, Turpie AGG, Verheugt FWA, Kakkar AK; GARFIELD-AF Investigators. Improved risk stratification of patients with atrial fibrillation: an integrated GARFIELD-AF tool for the prediction of mortality, stroke and bleed in patients with and without anticoagulation. BMJ Open. 2017 Dec 21;7(12):e017157. doi: 10.1136/bmjopen-2017-017157. PMID 29273652
- [Derived] Fox KAA, Accetta G, Pieper KS, Bassand JP, Camm AJ, Fitzmaurice DA, Kayani G, Kakkar AK; GARFIELD-AF Investigators. Why are outcomes different for registry patients enrolled prospectively and retrospectively? Insights from the global anticoagulant registry in the FIELD-Atrial Fibrillation (GARFIELD-AF). Eur Heart J Qual Care Clin Outcomes. 2018 Jan 1;4(1):27-35. doi: 10.1093/ehjqcco/qcx030. PMID 28950344
- [Derived] Camm AJ, Accetta G, Al Mahmeed W, Ambrosio G, Goldhaber SZ, Haas S, Jansky P, Kayani G, Misselwitz F, Oh S, Oto A, Raatikainen P, Steffel J, van Eickels M, Kakkar AK; GARFIELD-AF Investigators. Impact of gender on event rates at 1 year in patients with newly diagnosed non-valvular atrial fibrillation: contemporary perspective from the GARFIELD-AF registry. BMJ Open. 2017 Mar 6;7(3):e014579. doi: 10.1136/bmjopen-2016-014579. PMID 28264833
- [Derived] Haas S, Ten Cate H, Accetta G, Angchaisuksiri P, Bassand JP, Camm AJ, Corbalan R, Darius H, Fitzmaurice DA, Goldhaber SZ, Goto S, Jacobson B, Kayani G, Mantovani LG, Misselwitz F, Pieper K, Schellong SM, Stepinska J, Turpie AG, van Eickels M, Kakkar AK; GARFIELD-AF Investigators. Quality of Vitamin K Antagonist Control and 1-Year Outcomes in Patients with Atrial Fibrillation: A Global Perspective from the GARFIELD-AF Registry. PLoS One. 2016 Oct 28;11(10):e0164076. doi: 10.1371/journal.pone.0164076. eCollection 2016. PMID 27792741
- [Derived] Camm AJ, Accetta G, Ambrosio G, Atar D, Bassand JP, Berge E, Cools F, Fitzmaurice DA, Goldhaber SZ, Goto S, Haas S, Kayani G, Koretsune Y, Mantovani LG, Misselwitz F, Oh S, Turpie AG, Verheugt FW, Kakkar AK; GARFIELD-AF Investigators. Evolving antithrombotic treatment patterns for patients with newly diagnosed atrial fibrillation. Heart. 2017 Feb 15;103(4):307-314. doi: 10.1136/heartjnl-2016-309832. Epub 2016 Sep 19. PMID 27647168
- [Derived] Oh S, Goto S, Accetta G, Angchaisuksiri P, Camm AJ, Cools F, Haas S, Kayani G, Koretsune Y, Lim TW, Misselwitz F, van Eickels M, Kakkar AK; GARFIELD-AF Investigators. Vitamin K antagonist control in patients with atrial fibrillation in Asia compared with other regions of the world: Real-world data from the GARFIELD-AF registry. Int J Cardiol. 2016 Nov 15;223:543-547. doi: 10.1016/j.ijcard.2016.08.236. Epub 2016 Aug 13. PMID 27552578
- [Derived] Bassand JP, Accetta G, Camm AJ, Cools F, Fitzmaurice DA, Fox KA, Goldhaber SZ, Goto S, Haas S, Hacke W, Kayani G, Mantovani LG, Misselwitz F, Ten Cate H, Turpie AG, Verheugt FW, Kakkar AK; GARFIELD-AF Investigators. Two-year outcomes of patients with newly diagnosed atrial fibrillation: results from GARFIELD-AF. Eur Heart J. 2016 Oct 7;37(38):2882-2889. doi: 10.1093/eurheartj/ehw233. Epub 2016 Jun 29. PMID 27357359
- [Derived] Lip GY, Rushton-Smith SK, Goldhaber SZ, Fitzmaurice DA, Mantovani LG, Goto S, Haas S, Bassand JP, Camm AJ, Ambrosio G, Jansky P, Al Mahmeed W, Oh S, van Eickels M, Raatikainen P, Steffel J, Oto A, Kayani G, Accetta G, Kakkar AK; GARFIELD-AF Investigators. Does sex affect anticoagulant use for stroke prevention in nonvalvular atrial fibrillation? The prospective global anticoagulant registry in the FIELD-Atrial Fibrillation. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2 Suppl 1):S12-20. doi: 10.1161/CIRCOUTCOMES.114.001556. Epub 2015 Feb 24. PMID 25714828
- See also: Sponsor's website — http://www.tri-london.ac.uk/garfield